CLINICAL TRIAL: NCT04680624
Title: Role of Brodalumab in the Modulation of Gut Microbiome in Psoriatic Patient - BOMOGUMIP
Brief Title: Role of Brodalumab in the Modulation of Gut Microbiome in Psoriatic Patients
Acronym: BOMOGUMIP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Association pour la Recherche Clinique et Immunologique (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 20071A0005
Record Dates: First submitted 2020-12-11; First posted 2020-12-23 (Actual); Last update posted 2020-12-23 (Actual); Status verified 2020-12

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Group (Other)
  Interventions: Procedure: Fecal sample collection

INTERVENTIONS:
Procedure: Fecal sample collection — During the study, patients will be ask to collect fecal samples using sample collection kits. A total of 4 stool samples per patient will be collected.

SUMMARY:
BOMOGUMIP is an interventional research with minimal risk and constraints (cat.2), exploratory, intra-individual, prospective, multi-site study. The main objective of this intra individual prospective study is to determine the evolution of microbial composition of fecal samples issued to 15 patients after 6 months of Brodalumab treatment.

The population will consist of 15 adult patients suffering from moderate to severe skin psoriasis and starting, after having received a methotrexate treatment during at least 4 months, a brodalumab treatment in the first line of biological treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subject over 18 years of age
* Subject able to read, understand and give documented informed consent
* Subject willing and able to comply with the protocol requirements for the duration of the study
* Subject with health insurance coverage according to local regulations
* For woman with childbearing potential;

  * Use of a highly effective method of birth control from at least 1 month prior to study enrollment until the last visit
  * Negative urine pregnancy test at inclusion visit A highly effective method of birth controlled is defined as one which results in a low failure rate (i.e. less than 1% per year) when used consistently and correctly, such as implants, combined oral contraceptives, intrauterine device, barrier methods, sexual abstinence or vasectomized partner.

Woman with no childbearing potential is defined as: woman with amenorrhea for at least 12 months (without an alternative medical cause); woman who had undergone a permanent sterilization method (eg bilateral tubal occlusion which includes tubal ligation procedures, hysterectomy, bilateral salpingectomy, bilateral oophorectomy); or otherwise be incapable of pregnancy.

* Subject diagnosed with plaque psoriasis
* Subject treated with methotrexate (≥ 15mg/weeks) for at least 4 months and having inadequate response or intolerance to methotrexate treatment
* Subject starting a Brodalumab treatment as a first line of biological treatment (switching from methotrexate to Brodalumab treatment) Note: treatment decision must has been taken by the investigator prior to, and independently of the patient inclusion into the study. Thus, all recommendation and contraindication to the use of Brodalumab will be applicable (see section 6. Treatment).

Exclusion Criteria:

* Pregnancy or breast-feeding women, or planning to change contraception method or become pregnant or breastfeed during the study
* Subject currently experiencing or having a history of other concomitant skin conditions that would interfere with evaluation of psoriasis
* Subject treated by immunosuppressant drug except methotrexate (e.g. phototherapy, ciclosporin, apremilast, steroids or other systemic immunosuppressive) within 3 months before inclusion
* Subject treated by Non-Steroidal Anti-Inflammatory Drugs (NSAID), antibiotics or proton-pump inhibitors within 4 weeks before inclusion or foreseeable use during the study
* Subject previously treated by a biologic therapy
* Subject with a concomitant diagnosis of cirrhosis, coeliac disease or sign of bacterial infection
* Subject having a personal or familial history of psoriatic arthritis or inflammatory bowel disease
* Subject with a Body Mass Index (BMI)<18.5 or BMI>35
* Subject consuming probiotics or using specific diet (e.g. gluten-free, vegetarian, vegan, intermittent fasting) or planning to adopt a specific diet during the study
* Subject having a planned surgery during the study
* Subject presenting clinically significant medical disease that is uncontrolled despite treatment that is likely, in the opinion of the investigator, to impact patient's ability to participate in the study or to impact the study efficacy or safety assessments
* Subject with any additional condition that, in the opinion of the investigator, may interfere with the assessment or put the subject at risk
* Linguistic or mentally incapacity to sign the consent form
* Subject protect by the law (adult under guardianship, or hospitalized in a public or private institution for a reason other than study, or incarcerated)
* Subject in an exclusion period from a previous study or who is participating in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Evolution of microbial composition of fecal samples after 6 months of Brodalumab treatment. | At 6 months (Comparison V3/V1)
  Microbial features impacted by anti-interleukin-17 treatment (Brodalumab).